CLINICAL TRIAL: NCT03697226
Title: An Open-Label Multiple-Dose, Dose Escalation Study To Evaluate Safety, Tolerability and Pharmacokinetics of Topical ABI-1968 in Participants With Cervical High Grade Squamous Intraepithelial Lesions
Brief Title: Study of Topical ABI-1968 in Subjects With Precancerous Cervical Lesions From Human Papillomavirus (HPV) Infection.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Antiva Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ABI-1968-103
Record Dates: First submitted 2018-09-25; First posted 2018-10-05 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2019-07

CONDITIONS: HSIL of Cervix; HSIL, High Grade Squamous Intraepithelial Lesions; High-Grade Cervical Intraepithelial Neoplasia; Human Papilloma Virus; HIV Negative; Cervical Cancer; CIN - Cervical Intraepithelial Neoplasia; Cervical Neoplasm; Cervical Dysplasia
MeSH Terms: conditions — Squamous Intraepithelial Lesions; Uterine Cervical Neoplasms; Uterine Cervical Dysplasia

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose 1 (Experimental): Topical ABI-1968 Cream applied at Day 1, Day 8, Day 15 and Day 22
  Interventions: Drug: Topical ABI-1968
- Dose 2 (Experimental): Topical ABI-1968 Cream applied at Day 1, Day 8, Day 15 and Day 22
  Interventions: Drug: Topical ABI-1968
- Dose 3 (Experimental): New Topical ABI-1968 Formulation applied at Day 1, Day 8, Day 15 and Day 22
  Interventions: Drug: Topical ABI-1968
- Dose 4 (Experimental): New Topical ABI-1968 Formulation applied at Day 1, Day 8, Day 15 and Day 22
  Interventions: Drug: Topical ABI-1968
- Dose 5 (Experimental): New Topical ABI-1968 Formulation applied at Day 1, Day 8, Day 15 and Day 22
  Interventions: Drug: Topical ABI-1968

INTERVENTIONS:
Drug: Topical ABI-1968 — Multiple Doses of Topical ABI-1968 Cream with 4 once weekly doses administered in up to 5 Cohorts

SUMMARY:
This study evaluates the use of ABI-1968, a topical cream, in the treatment of cervical precancerous lesions in females without human immunodeficiency virus (HIV) infection.

ELIGIBILITY:
Inclusion Criteria:

1. Women, 25 to 50 years old.
2. Biopsy-confirmed cervical HSIL that is p16+ within 60 days of enrollment (dosing) with no evidence of invasive cancer in any specimen.
3. Colposcopy is satisfactory based on visualization of the entire squamo-columnar junction (SCJ). The borders of all lesions must be completely visible.
4. The upper limit of the visible (usually aceto-white) lesion is within 3 quadrants or less at screening.

Exclusion Criteria:

1. Women who are pregnant, plan to become pregnant in the next 4 months, or lactating females.
2. HIV positive (tested at screening visit or within 3 months of screening visit).
3. Resolution of visible CIN lesion prior to enrollment.
4. ECC positive for glandular disease (adenocarcinoma in situ) or invasive cancer.
5. History of cervical cancer, colposcopy suspicious for cancer, any prior treatment of CIN, or hysterectomy.

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 8 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2020-05-26 (Actual); Study Completion 2020-06-12 (Actual)

PRIMARY OUTCOMES:
Safety & Tolerability of ABI-1968 for the treatment of cHSIL | 42 days
  Number of Adverse Events related to treatment

SECONDARY OUTCOMES:
Systemic exposure to ABI-1968 Topical Cream following topical application to the cervix. | 42 days
  Plasma concentrations of ABI-1968 over time

OTHER OUTCOMES:
Histopathology of areas with biopsy-proven disease | 42 days
  Number of subjects with complete and or partial regression of cHSIL by Histopathology
Changes in HPV viral load following multiple doses of ABI-1968 Topical Cream | 42 days
  Changes from baseline in HPV viral load following multiple doses of ABI-1968 Topical Cream

CONTACTS AND LOCATIONS:
Locations (1):
- Research Center, Bloemfontein, Free State, South Africa

IPD SHARING:
Plan to Share IPD: No